CLINICAL TRIAL: NCT03374969
Title: Differential DNA Methylation as a Function of a Parenting Intervention: A Randomized Clinical Trial
Brief Title: Differential DNA Methylation as a Function of a Parenting Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Delaware (Other)
Responsible Party: Principal Investigator, Mary Dozier, Professor, Unidel Amy Elizabeth du Pont Chair in Child Development, Director of Clinical Training, University of Delaware
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 511457
Record Dates: First submitted 2017-12-12; First posted 2017-12-15 (Actual); Last update posted 2017-12-19 (Actual); Status verified 2017-12

CONDITIONS: Maltreatment, Child

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Attachment and Biobehavioral Catch-Up (Experimental)
  Interventions: Behavioral: Attachment and Biobehavioral Catch-Up
- Developmental Education for Families (Active Comparator)
  Interventions: Behavioral: Developmental Education for Families

INTERVENTIONS:
Behavioral: Attachment and Biobehavioral Catch-Up — Attachment and Biobehavioral Catch-up (ABC) is a 10-session, weekly intervention delivered in the family's home. ABC addresses three primary issues. First, young children who have experienced early adversity are especially in need of nurturance and parents who behave in synchronous ways and delight in them. Next, when parents behave in frightening ways, it is difficult for children to look to them for reassurance when distressed. This can be particularly difficult for children who have experienced early adversity. Therefore, this intervention helps parents learn how to: 1) behave in nurturing ways when children are distressed; 2) behave in synchronous, delighted ways when children are not distressed; and 3) avoid behaving in frightening or intrusive ways. Interventionists are provided with a manualized protocol, but tailor specific session content to each family's needs. Sessions are videotaped, both for playback to families, and for supervision.
  Arms: Attachment and Biobehavioral Catch-Up
Behavioral: Developmental Education for Families — Developmental Education for Families (DEF) is a 10-session, weekly intervention delivered in the family's home. DEF focuses on enhancing gross and fine motor skills, cognition and language development. The age-based protocols (i.e., 6-24 months,) provide information about the developmental themes of focus for each week and suggest activities to enhance the target skills for that week. However, the protocols do not provide a direct script with which to conduct the sessions. Interventionists tailor the developmental program session to the needs of the child and family by considering the child's current gross, fine, cognitive and language skills and creatively preparing several activities that will address the session topics.
  Arms: Developmental Education for Families

SUMMARY:
The aim of this study is to experimentally assess whether an early parenting intervention for maltreating parents results in differential epigenetic marking of children's genome, particularly of DNA associated with immune system functioning, obesity, and mental health.

DETAILED DESCRIPTION:
This study assesses whether a 10-session intervention for maltreating parents effects the epigenome of young children who have experienced early maltreatment. Families are randomly assigned to the experimental condition (Attachment and Biobehavioral Catch-Up) or a treatment control (Developmental Education for Families). Biological samples and behavioral observations of parenting will be collected pre- and post- intervention. Biological samples will be used to conduct whole genome analyses of differential DNA methylation that occur as a result of the intervention. Behavioral observations of parent-child interactions will be used to assess the efficacy of the intervention in altering parenting behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Parents will be considered potentially eligible if they have a child between the ages of 6 and 20 months and have a history of substantiated or unsubstantiated report of maltreatment or domestic violence. After obtaining informed consent, observational assessments of sensitivity will be conducted, allowing screening of parents with low levels of sensitivity (who are expected to benefit more from the intervention than others). Only those parents who have scores in the insensitive range will be included in the full study.

Exclusion Criteria:

* Children with known serious medical issues (e.g., cerebral palsy) will be excluded from the sample. Also, high-risk parents will be screened for sensitivity to ensure that they will benefit from the intervention. Only those who are screened as relatively insensitive (1-2 on a 5 point coding scale) will be included in the full study.
* If the primary caregiver loses custody of the child before completion of the project, the participant will be withdrawn from the study.
* If the primary caregiver is incarcerated before completion of the study, the subject will be withdrawn from the study.

Ages: 6 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2013-12-09 (Actual); Primary Completion 2014-12-16 (Actual); Study Completion 2017-02-10 (Actual)

PRIMARY OUTCOMES:
Whole Genome DNA Methylation | from date of enrollment to 1 month after completing the intervention

SECONDARY OUTCOMES:
Parental Sensitivity | On date of enrollment, each intervention session, and 1 month after completing the intervention